CLINICAL TRIAL: NCT06926933
Title: An Open Label, Single-group, Multicenter Study on the Efficacy and Safety of Leuprolide Acetate 45 mg for Injectable Suspension-controlled Release in Subjects With Central (Gonadotropin-dependent) Precocious Puberty
Brief Title: Efficacy and Safety of Leuprolide Acetate 45 mg in Subjects With Central Precocious Puberty
Acronym: NEST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLA24IV_1
Record Dates: First submitted 2025-04-08; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: CPP
MeSH Terms: interventions — luprolide acetate gel depot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eligard® 45 mg (Experimental): SC injection of study drug (45 mg of leuprolide acetate for injectable suspensions)
  Interventions: Drug: Eligard® 45 mg

INTERVENTIONS:
Drug: Eligard® 45 mg — 45 mg of leuprolide acetate

SUMMARY:
This study is a multicenter, open-label, single-group, and phase 4 study to evaluate the efficacy and safety of 45 mg of leuprolide acetate in CPP.

Screening tests are performed after the subject agrees in writing to participate in the clinical trial, and subjects who meet the inclusion criteria and do not fall under the exclusion criteria are enrolled in the study. The target patients in this study are pediatric patients who have been diagnosed with CPP but have not yet received GnRH agonist treatment, and all subjects perform GnRH stimulation tests to confirm their CPP diagnosis.

ELIGIBILITY:
Inclusion Criteria:

1. Pubertal-type LH response following an abbreviated GnRH stimulation test before treatment initiation > 5 IU/L
2. A subject manifested with central precocious puberty according to the following criteria Age : Boy (4 years of age or older ~ under 9 years of age) Girl (4 years of age or older ~ under 8 years of age) Tanner Stage : Level 2 or higher
3. Based on baseline visit (Day 0), those under the age of 10 for boys and those under the age of 9 for girls
4. Confirmed diagnosis of CPP within 12 months of Baseline Visit (Day 0) but have not received prior GnRH agonist treatment for CPP
5. Children with a body weight of more than 20 kg at screening
6. Children have a bone age that is ≥1 year older than their chronological age at screening
7. A signed written consent form by a legal representative who has been informed about this study

Exclusion Criteria:

1. Gonadotropin-independent (peripheral) precocious puberty: extra pituitary secretion of gonadotropins or gonadotropin-independent gonadal or adrenal sex steroid secretion
2. Prior or current GnRH treatment for CPP
3. Non-progressing isolated premature thelarche
4. Presence of an unstable intracranial tumor or an intracranial tumor requiring neurosurgery or cerebral irradiation. Subjects with hamartomas not requiring surgery are eligible.
5. Prior (within 12 weeks of Screening) use of medications

   * Hormonal agonists (Estrogen, Progesterone, FSH, LH, Testosterone etc.)
   * Hormonal antagonists (Anti-Estrogen agents, Anti-Androgen agents)
   * Steroid use (except for mild topical steroids, oral steroids are allowed within 30 days)
   * Herbal Medicines
6. Prior or current therapy with growth hormone
7. Major medical or psychiatric illness that could interfere with study visits
8. Diagnosis of short stature (i.e. 2 standard deviations (SD) below the mean height for age or 3rd percentile for age)
9. Pregnant or likely pregnant women (Positive urine pregnancy test), nursing women
10. Known hypersensitivity to GnRH or related compounds
11. Any other medical condition or serious intercurrent illness that, in the opinion of the investigator, may make it undesirable for the subject to participate in the study
12. Any other condition(s) which could significantly interfere with Protocol compliance
13. Treatment with an investigational product within 5 half-lives of that product in prior clinical studies before the baseline visit (Day 0)
14. Known history of seizures, epilepsy, and/or central nervous system disorders that may be associated with seizures or convulsions
15. Prior (within 6 months of Baseline (Day 0)) or current use of medications that, per investigator opinion, have been associated with seizures or convulsions

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
The percentage (%) of subjects with serum LH concentrations < 4 IU/L following an GnRH stimulation test | at week 24
  Blood samples for serum LH concentrations (as appropriate) will be collected at the appropriate assessment times and analyzed by a central laboratory.

SECONDARY OUTCOMES:
The percentage (%) of subjects with suppressed serum LH concentrations (< 4 IU/L) 30-minutes post GnRH stimulation test | at week 12, 48, 72, 96
  Blood samples for serum LH concentrations (as appropriate) will be collected at the appropriate assessment times and analyzed by a central laboratory.
The percentage (%) of subjects with suppressed serum FSH (< 2.5 mIU/mL), estradiol (< 20 pg/mL, for girl) or testosterone (< 30 ng/dL, for boy) | at week 12, 24, 48, 72, 96
  Sexual development in puberty will be assessed by Tanner staging
The percentage of subject of Tanner stage (including menstruation) | at week 12, 24, 48, 72, 96
  Sexual development in puberty will be assessed by Tanner staging
Height velocity (growth rate) | at week 12, 24, 48, 72, 96
  Annualized Height Velocity
The ratio of bone age and chronological age | at week 12, 24, 48, 72, 96
  A single X-ray of the non-dominant hand and wrist will be obtained periodically

CONTACTS AND LOCATIONS:
Overall Officials: Eunhee Lee, Study Director — Hanall Biopharma
Locations (9):
- South Korea (9):
  - Korea University Ansan Hospital, Ansan
  - Jeonbuk National University Hospital, Jeonju
  - Chosun University Hospital, Kwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Kyung Hee University Hospital At Gangdong, Seoul
  - Ajou University Medical Center, Suwon